CLINICAL TRIAL: NCT06230185
Title: Breast Cancer-Minimal/Molecular Residual Disease Detection and Therapy Monitoring in Patients with Early Stage TNBC-Phase I (B-STRONGER-I)
Brief Title: CtDNA Based MRD Testing for NAC Monitoring in TNBC
Acronym: B-STRONGER-I
Status: Recruiting | Type: Observational
Sponsor: Personalis Inc. (Industry)
Responsible Party: Principal Investigator, Pavani Chalasani, Director, Division of Hematology and Oncology, George Washington University
Other Study IDs: 01-PS-001; B-STRONGER-I (Other: Personalis)
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: TNBC - Triple-Negative Breast Cancer; Minimal Residual Disease
Keywords: ctDNA; Liquid Biopsy; Breast Cancer; MRD; NAC; TNBC; NeXT Personal®
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm, Residual; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE, DNA extracted from blood, ctDNA extracted from plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A prospective, multicenter, observational study to evaluate the correlation of Molecular Residual Disease (MRD) detection using circulating tumor DNA guided test to pathological complete response (pCR) after neoadjuvant chemotherapy (NAC) in stage I-III triple negative breast cancer (TNBC). Results from this study aim to improve MRD detection and disease outcomes for future patients.

DETAILED DESCRIPTION:
NeXT Personal CTA (Clinical Trial Assay) is a patient-specific, tumor-informed device which allows for detection of MRD from cfDNA. By using next generation sequencing technology, whole genome sequencing (WGS) is conducted from DNA derived from patient tumor and normal samples. A tumor informed personalized panel is then constructed that uses only a selection of DNA targets from the WGS by applying bioinformatic filters. The targeted personalized panel is then sequenced using NGS and DNA derived from cfDNA from plasma samples. The data from the cfDNA NGS are then further analyzed using bioinformatics filters to report the MRD status.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically documented TNBC (defined as ER expression ≤10% by IHC, PR expression≤10% by IHC and HER2 0 or 1+ by IHC or FISH ratio <2 or HER2 gene copy number of <6).
2. Early-stage breast cancer (stage I-III) and scheduled to undergo NAC treatment with curative intent.
3. Be informed of the investigational nature of the study and all pertinent aspects of the trial.
4. Have the ability to understand and the willingness to sign a written informed consent document in accordance with institutional and federal guidelines.
5. Be ≥ 18years of age.
6. Patient who are scheduled to start NAC.
7. Be willing to provide blood samples before and during treatment.
8. Have available biopsy tissue.

Exclusion Criteria:

1. Receiving concurrent anti-neoplastic therapy for another malignancy.
2. Stage IV disease.
3. Current or history of another primary cancer within 5 years of study entry, with the exception of basal or squamous cell skin cancer, or non-invasive malignancy.
4. History of allogeneic bone marrow or organ transplant.
5. Blood transfusion within two weeks before collection of blood for central ctDNA testing.
6. Started systemic therapy for their breast cancer.
7. Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patient who are scheduled to start NAC with early-stage Triple Negative Breast Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 422 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the correlation of MRD to pCR after NAC in TNBC | through study completion, an average of 6 months
  Evaluate the correlation of MRD detection by NeXT Personal CTA to pathological Complete Response (pCR) after neoadjuvant chemotherapy (NAC) in stage I-III triple negative breast cancer (TNBC). The pCR is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy.

SECONDARY OUTCOMES:
Evaluate the trajectory of changes in MRD to pCR or non pCR in TNBC | through study completion, an average of 6 months
  Evaluate the trajectory of changes in MRD detected by NeXT Personal CTA during neoadjuvant chemotherapy (NAC) to pathological Complete Response (pCR) or non pCR in stage I-III triple negative breast cancer (TNBC).

OTHER OUTCOMES:
Stratification based on NAC therapy regimen | through study completion, an average of 6 months
  NeXT Personal CTA clinical accuracy may be evaluated as compared to other clinically available tests. Stratification based on NAC therapy regimen, genomic profiles and biomarker analysis.
Evaluate genomic profiles | through study completion, an average of 6 months
  Evaluate genomic profile for specific biomarkers during neoadjuvant chemotherapy (NAC)

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, Principal Investigator — George Washington University
Locations (14):
- United States (14):
  - Arizona Oncology, Tucson, Arizona
  - University of Colorado Cancer Center, Aurora, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Mount Sinai Medical Center of Florida, Miami Beach, Florida
  - Comprehensive Hematology Oncology (ONare Alliance, LLC / Exigent Research, LLC, St. Petersburg, Florida
  - Illinois Cancer Care, Peoria, Illinois
  - Louisiana State University, New Orleans, Louisiana
  - Trinity Health-Michigan, Ypsilanti, Michigan
  - Nebraska Methodist, Omaha, Nebraska
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Oregon Oncology Specialists, Salem, Oregon
  - Cancer Care Associates of York, York, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Northwest, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided